CLINICAL TRIAL: NCT04513041
Title: Comparison of Pinhole Surgical Technique and Tunnel Technique for the Treatment of Gingival Recession: A Split Mouth Clinical and Digital Study
Brief Title: Pinhole Versus Tunnel for Soft Tissue Recession
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohanad Al-Sabbagh (Other)
Responsible Party: Sponsor-Investigator, Mohanad Al-Sabbagh, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80275
Record Dates: First submitted 2020-07-29; First posted 2020-08-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Right and left sides of the mouth will be randomly assigned to test and control group by computer generated randomization table in a split mouth design
Masking Description: PI and statistician will be blinded to the type of investigation for
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pinhole/Tunnel (Experimental): Participants will receive Pinhole surgical technique for treatment of soft tissue recession at one side of the mouth and Tunnel technique for treatment of soft tissue recession at the other side of the mouth
  Interventions: Procedure: Pinhole surgical technique and tunnel technique in a split mouth design

INTERVENTIONS:
Procedure: Pinhole surgical technique and tunnel technique in a split mouth design — Each subject will have the each surgical procedure which are both considered routine minimally invasive clinical care for gingival recession. Gum recession on one side will receive Pinhole surgical technique (test procedure). The other side will receive Tunnel technique (control procedure), Research component involved is the capture of digital impression using intra-oral scanner in the baseline (preoperative) and the final visit (6 months postoperative).

SUMMARY:
This is an assessor-blinded split-mouth randomized clinical study to compare root coverage and gingival tissue thickness following two different surgical procedures for non-autologous grafting: the pinhole surgical technique (PST) and tunnel technique.

DETAILED DESCRIPTION:
Each patient will undergo both surgeries on either quadrant; the PST and tunnel technique. The site will be randomized to receive either type of surgeries. Both types of surgeries are considered minimally invasive procedures to obtain root coverage for gingival recession. Both surgeries are clinically utilized in clinical practice and yield comparable results according to the literature, however, No prospective studies are published to compare between the outcomes of both techniques. patients will receive intra oral scan before the surgery and 6 months after the surgery to compare change in root coverage and gingival thickness outcomes between the two techniques. Post operative pain as well as patient satisfaction will be measured by visual analog scale and compared between the two techniques. Patients will be monitored at different time points to asses healing.

ELIGIBILITY:
Inclusion Criteria:

* between 18-75 years old
* have at least one non-mobile tooth with Cairo class I gingival recession of 2 to 6 mm.
* American Society of Anesthesiology class I and II
* full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) below 20%

Exclusion Criteria:

* sites of gingival recession around teeth that are non-salvageable
* presence of any exudate, infection or local inflammation around the area to be grafted
* pregnant or breastfeeding females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in gingival thickness | 6 months (pre operative and at the 6-month follow-up visit)
  Two digital scans (pre- and 6-month post-operative) will be overlapped to measure the change in gingival thickness.
Change in gingival recession | 6 months (pre operative and at the 6-month follow-up visit)
  Two digital scans (pre- and 6-month post-operative) will be overlapped to measure the change in gingival recession.

SECONDARY OUTCOMES:
Change in papillary recession | 6 months (pre operative and at the 6-month follow-up visit)
  Two digital scans (pre- and 6-month post-operative) will be overlapped to measure papillary gingival recession.
Change in root coverage | 6 months (pre operative and at the 6-month follow-up visit)
  Two digital scans (pre- and 6-month post-operative) will be overlapped to measure the complete elimination of gingival recession.
Change in sulcus probing depth | 6 months (pre operative and at the 6-month follow-up visit)
  During a clinical exam, a sulcus will be used to measure the depth from the free gingival margin to the base of the sulcus pre- and 6-months post-operative.
Change in clinical attachment. | 6 months (pre operative and at the 6-month follow-up visit)
  Clinical attachment will be calculated during the pre- and post-operative clinical exam.
Change in zone of keratinized tissue | 6 months (pre operative and at the 6-month follow-up visit)
  During a clinical exam, the zone of keratinized tissue will be measured during the pre- and post-operative clinical exam.
Change in bleeding on probing. | 6 months (pre operative and at the 6-month follow-up visit)
  The presence or absense of bleeding during probing during will be noted during the pre- and post-operative clinical exam.
Post-operative pain | 1 week
  A Visual Analog Score for pain will be used to assess post-operative pain one week after surgery. Scores range from 0-10; higher scores indicate greater pain.
Aesthetic satisfaction | 1 day
  A Visual Analog Score for aesthetic satisfaction will be used to assess patient satisfaction 6 months after surgery. Scores range from 0-10; higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad Al-Sabbagh, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Individual participants data will not be shared, rather the accumulated data for all participants could be shared to eliminate identification of participants.